CLINICAL TRIAL: NCT05325931
Title: 1-Week Dispensing Evaluation of Kalifilcon A Daily Disposable Multifocal Contact Lenses Compared to Ultra for Presbyopia Contact Lenses
Brief Title: 1-Week Dispensing Evaluation of Kalifilcon A Daily Disposable Multifocal Compared to Ultra for Presbyopia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: ROC2-22-005
Record Dates: First submitted 2022-04-01; First posted 2022-04-13 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: Presbyopia
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- kalifilcon A Daily Disposable Multifocal (Experimental): kalifilcon A Daily Disposable Multifocal Low Add Power (LA) and High Add Power (HA)
  Interventions: Device: kalifilcon A Daily Disposable Multifocal
- samfilcon A for Presbyopia (Active Comparator): B+L ULTRA for Presbyopia Low Add Power (LA) and High Add Power (HA)
  Interventions: Device: samfilcon A for Presbyopia

INTERVENTIONS:
Device: kalifilcon A Daily Disposable Multifocal — kalifilcon A Daily Disposable Multifocal low add and high
  Arms: kalifilcon A Daily Disposable Multifocal
Device: samfilcon A for Presbyopia — Ultra for Presbyopia Low and High Add Contact Lenses
  Arms: samfilcon A for Presbyopia

SUMMARY:
Experienced soft contact lens wearing subjects will be enrolled in this 1-week, confirmatory, randomized, bilateral, 2-way crossover, double masked (subject and investigator), repeated measures, dispensing study. All subjects will be seen for a Screening/Dispensing Visit at which informed consent will be obtained and eligibility will be assessed. If subjects satisfy all eligibility criteria and none of the exclusion criteria, subjects will be fit and dispensed study lenses according to unique randomization schedules that will be provided to each Investigator If vision is unsatisfactory in the original dispensed lenses, additional lens powers may be trialed.

ELIGIBILITY:
Inclusion Criteria:

* Be 40 years or older on the date the Informed Consent Form (ICF) is signed and have the capacity to read, understand and provide written voluntary informed consent.
* Have physiologically normal anterior segments not exhibiting clinically significant biomicroscopy findings.
* Have no active ocular disease or allergic conjunctivitis.
* Not be using any topical ocular medications.
* Be willing and able to follow instructions.
* Have signed a statement of informed consent.

Exclusion Criteria:

* Participating in a conflicting study.
* Considered by the Investigator to not be a suitable candidate for participation.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-02-25 (Actual); Primary Completion 2022-03-28 (Actual); Study Completion 2022-03-28 (Actual)

PRIMARY OUTCOMES:
Visual Acuity | One week
  Mean Binocular logMAR Visual Acuity at Distance (6m)
Near Visual Acuity | One week
  Mean Binocular logMAR Visual Acuity at Near (40cm)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Steffen, Study Director — Bausch & Lomb Incorporated
Locations (1):
- Bausch site 1, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No